CLINICAL TRIAL: NCT00475410
Title: A Phase III Multicenter, Single Blind, Randomized, Comparative and add-on Clinical Trial, in Three Parallel Groups, to Evaluate Efficacy and Safety of a New Therapy With Adipose-derived Autologous Stem Cells for the Treatment of Complex Perianal Fistulas in Patients Without Inflammatory Bowel Disease
Brief Title: Efficacy and Safety of Adipose Stem Cells to Treat Complex Perianal Fistulas Not Associated to Crohn´s Disease
Acronym: FATT1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tigenix S.A.U. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Cx401/FATT1; 2006-003370-95 (Other: EMEA)
Record Dates: First submitted 2007-05-17; First posted 2007-05-21 (Estimated); Last update posted 2019-04-12 (Actual); Status verified 2019-04

CONDITIONS: Anal Fistula
Keywords: Autologous adipose-derived stem cells; Complex perianal fistula; Inflammatory Bowel Disease; Advanced cell therapy; Fibrin glue
MeSH Terms: conditions — Rectal Fistula; Inflammatory Bowel Diseases | interventions — Fibrin Tissue Adhesive

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- ASCs (Experimental)
  Interventions: Drug: ASCs (Cx401, company code)
- ASCs+fibrin glue (Experimental)
  Interventions: Drug: ASCs (Cx401, company code); Drug: Fibrin adhesive
- Fibrin glue (Active Comparator)
  Interventions: Drug: Fibrin adhesive

INTERVENTIONS:
Drug: ASCs (Cx401, company code) — Experimental: ASCs: Subjects will be treated with a dose of 20 million ASCs and evaluated after 12 weeks. If needed a second dose of 40 million ASCs will be applied then.
  Experimental: ASCs+fibrin glue: Subjects will be treated with a dose of 20 million ASCs plus fibrin glue and evaluated after 12 weeks. If needed a second dose of 40 million ASCs plus fibrin glue will be applied then.
  Arms: ASCs; ASCs+fibrin glue
Drug: Fibrin adhesive — Experimental: Fibrin glue: Subjects will be treated with a dose fibrin glue and evaluated after 12 weeks. If needed a second dose of fibrin glue will be applied then.
  Arms: ASCs+fibrin glue; Fibrin glue

SUMMARY:
Anal fistula is defined as an abnormal communication between the anal canal and the perianal skin. Adipose-derived stem cells are a new therapy for the closure of these fistulas. This study will test the safety and efficacy of ASCs (adipose stem cells) in the treatment of patients without Crohn´s disease.

DETAILED DESCRIPTION:
Perianal fistula accounts for 10% to 30% of coloproctological surgical procedures. Currently accepted conventional treatment is surgery intended to treat the tracts using different technical options. This surgery usually has a highly bothersome postoperative period and may involve two major complications: anal incontinence and recurrence. The biological properties of stem cells derived from adult tissues make them adequate candidates for the treatment of diseases in which tissues are damaged or the healing process is altered. This study will compare the efficacy of ASCs versus ASCs plus Fibrin adhesive versus Fibrin adhesive alone for closure of complex perianal fistulas not associated to Inflammatory Bowel Disease. Fistula closure is defined as absence of suppuration and re-epithelization of the external opening in the clinical evaluation and absence of collections >2 cm directly related to the fistula tract treated, as measured by MRI

ELIGIBILITY:
Inclusion Criteria:

1. Patient with a complex perianal fistula. A complex perianal fistula must meet one of the following:

   * No fistula tract is palpated under the perianal skin or tract parallel to the rectum on examination with a stylet.
   * Associated anal incontinence in transsphincteric fistulas.
   * Risk factors for anal incontinence.
   * At least one prior surgery for a fistulous disease.
   * Suprasphincteric tracts shown by an image test.
2. Women of childbearing age should have a negative serum or urine pregnancy test (sensitive to 25IU of hCG) and not be lactating before study entry. Both men and women should use adequate birth control methods as defined by the investigator.
3. Seton presence is allowed at the time of study entry and until cells (in groups receiving ASCs) or Fibrin adhesive are implanted.
4. No condition that may prevent the patient from following the study procedures until 26 weeks of follow-up are completed is foreseen.
5. Patient should give his/her signed, written informed consent. -

Exclusion Criteria:

1. Patient has been diagnosed with IBD
2. Patient has a rectovaginal fistula
3. Patient is pregnant or lactating woman
4. Patient has acute sepsis at the time of study entry
5. A liposuction to draw at least 100 cc of fat from the abdominal wall is not technically feasible.
6. Patient needs surgery in the perianal region for reasons other than fistulas
7. Presence of two or more complex perianal fistulas
8. Patient has collections > 2 cm in MRI. If such collections exist, the surgeon may perform a complete toilette of the area.
9. Patient is allergic to local anesthetics or Gadolinium (MRI contrast agent).
10. MRI is not technically feasible.
11. Patient has abused alcohol or other addictive substances within 6 months of study entry.
12. Patient has active or latent infection by HIV, HBV or HCV.
13. Patient has undergone major surgery or sustained a severe trauma, in the investigator's judgment, within 28 days of recruitment.
14. Patient is receiving or has received immunomodulatory treatment for reasons other than the fistula within 6 months of study entry.
15. Patient has a malignant tumour, except for basal or squamous cell carcinoma of the skin, or has a prior history of a malignant tumour, except if the tumour has been in remission for at least the past 5 years.

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Actual)
Dates: Start 2007-02; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Closure of fistulas defined as absence of suppuration and re-epithelization of the external opening and absence of collections>2 cm directly related to the fistula tract treated, as measured by MRI (healing) | weeks 1, 4, 12 and 24. Week 26 in patients with a second dose

SECONDARY OUTCOMES:
• Clinical complexity of fistula (complexity of fistula score) • Safety: Cumulative incidence of adverse effects. • Quality of life (SF-36 score) • Degree of anal incontinence (Wexner incontinence score) | weeks 1, 4, 12 and 24. Week 26 in patients with a second dose

CONTACTS AND LOCATIONS:
Overall Officials: Damian Garcia Olmo, Dr, Principal Investigator
Locations (10):
- Universitary Clinical Surgery, Mannheim, Germany
- Spain (8):
  - Lozano Blesa Clinical Hospital, Zaragoza, Aragon
  - Virgen Del Camino Hospital, Pamplona, Navarre
  - Mutua de Terrasa Hospital, Tarrasa, Tarragona
  - Gregorio Marañon University Hospital, Madrid
  - San Carlos Clinical Hospital, Madrid
  - 12 De Octubre University Hospital, Madrid
  - La Paz University Hospital, Madrid
  - Universitary General Hospital, Valencia
- John Radcliff Hospital, Oxford, Oxfordshire, United Kingdom

REFERENCES:
- [Result] Garcia-Olmo D, Garcia-Arranz M, Herreros D, Pascual I, Peiro C, Rodriguez-Montes JA. A phase I clinical trial of the treatment of Crohn's fistula by adipose mesenchymal stem cell transplantation. Dis Colon Rectum. 2005 Jul;48(7):1416-23. doi: 10.1007/s10350-005-0052-6. PMID 15933795
- [Result] Garcia-Olmo D, Garcia-Arranz M, Garcia LG, Cuellar ES, Blanco IF, Prianes LA, Montes JA, Pinto FL, Marcos DH, Garcia-Sancho L. Autologous stem cell transplantation for treatment of rectovaginal fistula in perianal Crohn's disease: a new cell-based therapy. Int J Colorectal Dis. 2003 Sep;18(5):451-4. doi: 10.1007/s00384-003-0490-3. Epub 2003 May 20. PMID 12756590
- [Derived] Herreros MD, Garcia-Arranz M, Guadalajara H, De-La-Quintana P, Garcia-Olmo D; FATT Collaborative Group. Autologous expanded adipose-derived stem cells for the treatment of complex cryptoglandular perianal fistulas: a phase III randomized clinical trial (FATT 1: fistula Advanced Therapy Trial 1) and long-term evaluation. Dis Colon Rectum. 2012 Jul;55(7):762-72. doi: 10.1097/DCR.0b013e318255364a. PMID 22706128